CLINICAL TRIAL: NCT01096511
Title: Clinical Effectiveness and Safety Study of Moxifloxacin i.v. in the Treatment of Complicated Intra-Abdominal Infection (cIAI)
Brief Title: Moxifloxacin i.v. in the Treatment of Complicated Intra-Abdominal Infection (cIAI)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare Pharceuticals Inc.
Other Study IDs: 14537; AX0910CN (Other: company internal)
Record Dates: First submitted 2010-03-11; First posted 2010-03-31 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Secondary Peritonitis; Abscess, Intra-Abdominal
Keywords: Moxifloxacin,; cIAI; non-interventional
MeSH Terms: conditions — Peritonitis; Abdominal Abscess | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — The treatment with Moxifloxacin 400 mg infusion should comply with the recommendations written in the local product information. The decision about the treatment with Moxifloxacin as well as the duration of treatment is solely up to the attending physician.

SUMMARY:
This study is a local, prospective, open-label, company-sponsored, non interventional, multi-center study. Patients documented must suffer from a cIAI and take at least one dose of Moxifloxacin infusion.The primary objective is to define the types of cIAI infections that require Moxifloxacin i.v. therapy in China.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age with a diagnosis of cIAI treated with Moxifloxacin infusion with/without sequential tablet treatment can be included into the study. The local Moxifloxacin product information must be considered.

Exclusion Criteria:

* Contraindications stated in the local Moxifloxacin product information. Warnings and precautions, stated in the local Moxifloxacin product information must be considered as potential exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients with cIAI, who are at least 18 years of age and are scheduled to be treated with Moxifloxacin infusion, can be documented after the therapy decision has been made.
Sampling Method: Non-Probability Sample
Enrollment: 1001 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Types of cIAI infections | Day 1

SECONDARY OUTCOMES:
Cure rate | 5-14 days
Clinical signs and symptoms | 5-14 days
Duration until improvement and cure | 5-14 days
Adverse event collection | 5-14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China